CLINICAL TRIAL: NCT04973449
Title: A Phase II/III Partially Double-Blinded, Randomised, Multinational, Active-Controlled Study in Both Previously Vaccinated and Unvaccinated Adults to Determine the Safety and Immunogenicity of AZD2816, a Vaccine for the Prevention of COVID-19 Caused by Variant Strains of SARS-CoV-2
Brief Title: Phase II/III Study of AZD2816, for the Prevention of COVID-19 in Adults
Acronym: AZD2816
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D7220C00001; 2021-002530-17 (EudraCT Number)
Record Dates: First submitted 2021-07-02; First posted 2021-07-22 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Intervention Model Description: Previously vaccinated individuals will receive 1 dose of
  AZD1222 or AZD2816 on Day 1. Previously unvaccinated participants will receive one of the following 2-dose vaccinations:
  * 1 dose of AZD2816 on Day 1 and on Day 29
  * 1 dose of AZD1222 on Day1 and on Day 29
  * 1 dose of AZD1222 on Day 1 and 1 dose of AZD2816 on Day 29
  * 1 dose of AZD2816 on Day 1 and on Day 85. Participants will be followed up for safety for 180 days after last study vaccine administration.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind: two or more parties are unaware of the intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Primary Vaccination Cohort:- AZD1222 (4) (Experimental): Previously unvaccinated participants received intramuscular (IM) AZD1222 5*10^10 viral particles (vp) on Days 1 and 29 (4-week dosing interval).
  Interventions: Biological: AZD1222
- Primary Vaccination Cohort:- AZD2816 (4) (Experimental): Previously unvaccinated participants received IM AZD2816 5*10^10 vp on Days 1 and 29 (4-week dosing interval).
  Interventions: Biological: AZD2816
- Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (Experimental): Previously unvaccinated participants received IM AZD1222 5*10^10 vp on Day 1 and IM AZD2816 5*10^10 vp on Day 29 (4-week dosing interval).
  Interventions: Biological: AZD1222; Biological: AZD2816
- Primary Vaccination Cohort:- AZD2816 (12) (Experimental): Previously unvaccinated participants received IM AZD2816 5*10^10 vp on Days 1 and 85 (12-week dosing interval).
  Interventions: Biological: AZD2816
- Booster Cohort:- AZD1222:AZD1222 (Experimental): Participants, who previously received 2 doses of AZD1222 vaccine according to the authorized dose and dosing regimen, with second dose administered at least 90 days prior to study treatment, received booster dose of IM AZD1222 5*10^10 vp on Day 1.
  Interventions: Biological: AZD1222
- Booster Cohort:- AZD1222:AZD2816 (Experimental): Participants, who previously received 2 doses of AZD1222 vaccine according to the authorized dose and dosing regimen, with second dose administered at least 90 days prior to study treatment, received booster dose of IM AZD2816 5*10^10 vp on Day 1.
  Interventions: Biological: AZD2816
- Booster Cohort:- mRNA:AZD1222 (Experimental): Participants, who previously received 2 doses of approved mRNA based vaccine according to the authorized dose and dosing regimen, with second dose administered at least 90 days prior to study treatment, received booster dose of IM AZD1222 5*10^10 vp on Day 1.
  Interventions: Biological: AZD1222
- Booster Cohort:- mRNA:AZD2816 (Experimental): Participants, who previously received 2 doses of approved mRNA based vaccine according to the authorized dose and dosing regimen, with second dose administered at least 90 days prior to study treatment, received booster dose of IM AZD2816 5*10^10 vp on Day 1.
  Interventions: Biological: AZD2816

INTERVENTIONS:
Biological: AZD1222 — 10 mM histidine/histidine hydrochloride, 7.5% (w/v) sucrose, 35 mM sodium chloride, 1 mM magnesium chloride, 0.1% (w/v) polysorbate 80, 0.1 mM edetate disodium, 0.5% (w/v) ethanol, at pH 6.6.
  Arms: Booster Cohort:- AZD1222:AZD1222; Booster Cohort:- mRNA:AZD1222; Primary Vaccination Cohort:- AZD1222 (4); Primary Vaccination Cohort:- AZD1222 + AZD2816 (4)
Biological: AZD2816 — 10 mM histidine/histidine hydrochloride, 7.5% (w/v) sucrose, 35 mM sodium chloride, 1 mM magnesium chloride, 0.1% (w/v) polysorbate 80, 0.1 mM edetate disodium, 0.5% (w/v) ethanol, at pH 6.6.
  Arms: Booster Cohort:- AZD1222:AZD2816; Booster Cohort:- mRNA:AZD2816; Primary Vaccination Cohort:- AZD1222 + AZD2816 (4); Primary Vaccination Cohort:- AZD2816 (12); Primary Vaccination Cohort:- AZD2816 (4)

SUMMARY:
The aim of the study is to assess the safety, and immunogenicity of AZD2816 for the prevention of coronavirus disease 2019 (COVID-19).

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the safety and characterize the immunogenicity of AZD2816; AstraZeneca's candidate chimpanzee adenovirus Ox1 (ChAdOx1) vector vaccine against severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) variant strain B.1.351.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, ≥ 18 years of age at the time of consent.

   For inclusion in the SARS-CoV-2 seronegative population:
2. No history of laboratory-confirmed SARS-CoV-2 infection (ie, no positive nucleic acid amplification test and no positive antibody test).
3. Seronegative for SARS-CoV-2 at screening (lateral flow test to detect reactivity to the nucleoprotein).
4. Medically stable such that, according to the judgment of the investigator, hospitalization within the study period is not anticipated and the participant appears likely to be able to remain on study through the end of protocol-specified follow-up.
5. Able to understand and comply with study requirements/procedures (if applicable, with assistance by caregiver, surrogate, or legally authorized representative) based on the assessment of the investigator.
6. Signed informed consent obtained before conducting any study-related procedures.
7. Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   Previously COVID-19 Vaccinated Participants:
8. Prior completion of a 2-dose primary homologous vaccination regimen against SARSCoV-2 with either AZD1222 (2 standard doses as authorized vaccine or as investigational product in a clinical trial with a 4 to 12-week dosing interval) or with an mRNA vaccine approved for emergency or conditional use. The second dose in all cases should have been administered at least 3 months prior to first administration of study intervention.

Exclusion Criteria:

1. History of allergy to any component of AZD1222/AZD2816.
2. History of Guillain-Barré syndrome, any demyelinating disease, or any other neuroimmunologic condition.
3. Significant infection or other acute illness, including fever > 100 °F (> 37.8 °C) on the day prior to or day of randomization.
4. Any confirmed or suspected immunosuppressive or immunodeficient state, including asplenia or human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS).
5. Recurrent severe infections and use of immunosuppressant medication within the past 6 months (≥ 20 mg per day of prednisone or its equivalent, given daily or on alternate days for ≥ 15 days within 30 days prior to administration of study intervention). The following exceptions are permitted: Topical/inhaled steroids or short-term oral steroids (course lasting ≤ 14 days).
6. History of primary malignancy (see protocol).
7. History of thrombocytopenia and/or thrombosis, including participants who have experienced major venous and/or arterial thrombosis in combination with thrombocytopenia following vaccination with any COVID-19 vaccine.
8. History of heparin-induced thrombocytopenia, congenital thrombophilia (ie, factor V Leiden, prothrombin G20210A, antithrombin III deficiency, protein C deficiency and protein S deficiency, factor XIII mutation, familial dysfibrinogenemia), auto-immune thrombophilia (antiphospholipid syndrome, anti-cardiolipin antibodies, anti-β2- glycoprotein 1 antibodies), or paroxysmal nocturnal haemoglobinuria.
9. Clinically significant bleeding (eg, factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venepuncture.
10. Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, or neurological illness, as judged by the Investigator.
11. Any other significant disease, disorder, or finding that may significantly increase the risk to the participant because of participation in the study, affect the ability of the participant to participate in the study, or impair interpretation of the study data.
12. Any autoimmune conditions, except mild psoriasis and vitiligo.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2843 (Actual)
Dates: Start 2021-06-27 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- Brazil (5):
  - Research Site, Brasília
  - Research Site, Curitiba
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Salvador
- Poland (4):
  - Research Site, Lublin
  - Research Site, Oświęcim
  - Research Site, Puławy
  - Research Site, Zamość
- South Africa (4):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Somerset West
- United Kingdom (15):
  - Research Site, Birmingham
  - Research Site, Bournemouth
  - Research Site, Bristol
  - Research Site, Edinburgh
  - Research Site, Harrow
  - Research Site, Hull
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Nottingham
  - Research Site, Oxford
  - Research Site, Plymouth
  - Research Site, Portsmouth
  - Research Site, Sheffield
  - Research Site, Truro

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  URL:
  https://astrazenecagroup-dt.pharmacm.com/DT/Home
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Costa Clemens SA, Jepson B, Bhorat QE, Ahmad A, Akhund T, Aley PK, Bansal H, Bibi S, Kelly EJ, Khan M, Lambe T, Lombaard JJ, Matthews S, Pipolo Milan E, Olsson U, Ramasamy MN, Moura de Oliveira Paiva MS, Seegobin S, Shoemaker K, Szylak A, Villafana T, Pollard AJ, Green JA; AZD2816 Study Group. Immunogenicity and safety of beta variant COVID-19 vaccine AZD2816 and AZD1222 (ChAdOx1 nCoV-19) as primary-series vaccination for previously unvaccinated adults in Brazil, South Africa, Poland, and the UK: a randomised, partly double-blinded, phase 2/3 non-inferiority immunobridging study. Lancet Microbe. 2024 Aug;5(8):100863. doi: 10.1016/S2666-5247(24)00078-8. Epub 2024 Jun 12. PMID 38878794
- [Derived] Ramasamy MN, Kelly EJ, Seegobin S, Dargan PI, Payne R, Libri V, Adam M, Aley PK, Martinez-Alier N, Church A, Jepson B, Khan M, Matthews S, Townsend GT, Vekemans J, Bibi S, Swanson PA 2nd, Lambe T, Pangalos MN, Villafana T, Pollard AJ, Green JA; AZD2816 Study Group. Immunogenicity and safety of AZD2816, a beta (B.1.351) variant COVID-19 vaccine, and AZD1222 (ChAdOx1 nCoV-19) as third-dose boosters for previously vaccinated adults: a multicentre, randomised, partly double-blinded, phase 2/3 non-inferiority immunobridging study in the UK and Poland. Lancet Microbe. 2023 Nov;4(11):e863-e874. doi: 10.1016/S2666-5247(23)00177-5. Epub 2023 Sep 29. PMID 37783221
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7220C00001&attachmentIdentifier=0a3a6e16-16b7-4123-a7e4-f72724ff24f2&fileName=d7220c00001-sap-Redacted-27Jan23.pdf&versionIdentifier=
- See also: Clinical Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7220C00001&attachmentIdentifier=2702b48f-fd68-4497-ab85-0d17d2b22b0f&fileName=d7220c00001-16-1-01-protocol-and-protocol-amendments-final.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7220C00001&attachmentIdentifier=e750a312-5649-468d-b51e-8baf87ab2ae1&fileName=d7220c00001-final-synopsis-Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2843 participants were randomized in this study of which 2834 participants were treated (9 participants were randomized but not treated). Results are presented for 2834 treated participants only.
Period: Overall Study
Arm/Group | Primary Vaccination Cohort:- AZD1222 (4) | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD2816 (12) | Booster Cohort:- AZD1222:AZD1222 | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- mRNA:AZD1222 | Booster Cohort:- mRNA:AZD2816
Started | 409 | 413 | 411 | 208 | 373 | 377 | 322 | 321
Completed | 389 | 393 | 391 | 189 | 359 | 366 | 303 | 308
Not Completed | 20 | 20 | 20 | 19 | 14 | 11 | 19 | 13
Not completed — Withdrawal by Subject | 3 | 3 | 2 | 5 | 5 | 4 | 7 | 5
Not completed — Lost to Follow-up | 15 | 16 | 16 | 13 | 5 | 6 | 10 | 6
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 1 | 1 | 2 | 1 | 4 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomised participants who received study treatment, irrespective of their protocol adherence and continued participation in the study. Participants were analysed according to their randomised treatment assignment, irrespective of the treatment actually received.
Groups:
- Primary Vaccination Cohort:- AZD1222 (4): Previously unvaccinated participants received IM AZD1222 5*10^10 vp on Days 1 and 29 (4-week dosing interval).
- Total: Total of all reporting groups
Arm/Group | Primary Vaccination Cohort:- AZD1222 (4) | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD2816 (12) | Booster Cohort:- AZD1222:AZD1222 | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- mRNA:AZD1222 | Booster Cohort:- mRNA:AZD2816 | Total
Number analyzed (Participants) | 409 | 413 | 411 | 208 | 373 | 377 | 322 | 321 | 2834
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.1 (12.48) | 29.7 (12.95) | 28.0 (12.23) | 28.8 (12.98) | 59.7 (13.72) | 60.4 (13.30) | 55.3 (13.19) | 55.9 (13.73) | 43.2 (19.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 169 | 166 | 85 | 172 | 172 | 197 | 192 | 1324
  Male | 238 | 244 | 245 | 123 | 201 | 205 | 125 | 129 | 1510
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 239 | 246 | 257 | 131 | 8 | 10 | 4 | 6 | 901
  Not Hispanic or Latino | 143 | 148 | 137 | 70 | 322 | 331 | 291 | 292 | 1734
  Unknown or Not Reported | 27 | 19 | 17 | 7 | 43 | 36 | 27 | 23 | 199
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 8
  Asian | 3 | 5 | 4 | 0 | 10 | 14 | 8 | 13 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 202 | 192 | 214 | 98 | 2 | 1 | 3 | 2 | 714
  White | 161 | 166 | 151 | 86 | 325 | 328 | 290 | 288 | 1795
  More than one race | 11 | 23 | 10 | 6 | 0 | 1 | 2 | 0 | 53
  Unknown or Not Reported | 28 | 27 | 30 | 16 | 36 | 33 | 19 | 18 | 207

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local and Systemic Solicited Treatment Emergent Adverse Events (TEAEs) in Primary Vaccination Cohort (PVC):- AZD2816 (4), Booster Cohorts:-AZD1222:AZD2816, and mRNA:AZD2816
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. Solicited AEs are local or systemic predefined events for assessment of reactogenicity. An e-diary was used to collect information on the timing and severity of the solicited AEs. Local AEs included pain, redness/erythema, tenderness, induration/swelling at the site of the injection. Systemic AEs included fever (> 100 °F/37.8 °C), chills, muscle pains, fatigue, headache, malaise, nausea, and vomiting.
Time Frame: During the 7-day follow-up period after vaccination (vaccines administered on Days 1 and 29 [only for primary vaccination cohort])
Population: Seronegative safety analysis set included all participants who received at least 1 dose of study treatment, were analysed according to treatment actually received, and were seronegative at baseline. Here, number of participants analyzed denotes those participants who were evaluated for solicited symptoms.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Vaccination Cohort:- AZD2816 (4): Previously unvaccinated seronegative participants received IM AZD2816 5*10^10 vp on Days 1 and 29 (4-week dosing interval).
- Booster Cohort:- AZD1222:AZD2816: Seronegative participants, who previously received 2 doses of AZD1222 vaccine according to the authorized dose and dosing regimen, with second dose administered at least 90 days prior to study treatment, received booster dose of IM AZD2816 5*10^10 vp on Day 1.
- Booster Cohort:- mRNA:AZD2816: Seronegative participants, who previously received 2 doses of approved mRNA based vaccine according to the authorized dose and dosing regimen, with second dose administered at least 90 days prior to study treatment, received booster dose of IM AZD2816 5*10^10 vp on Day 1.
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- mRNA:AZD2816
Number analyzed (Participants) | 375 | 343 | 299
Participants
  Any solicited AEs | 319 | 275 | 277
  Any local solicited AEs | 278 | 225 | 236
  Any systemic solicited AEs | 289 | 211 | 253

2. Primary Outcome: Number of Participants With Unsolicited TEAEs, Treatment-emergent Serious AEs (TESAEs), Medically Attended AEs (MAAEs), and Adverse Events of Special Interest (AESIs) in PVC:- AZD2816 (4), Booster Cohorts:- AZD1222:AZD2816, and mRNA:AZD2816
Description: The AEs other than solicited AEs are reported as unsolicited AEs and were collected by "open question" at study visits. AE: any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. TEAEs: events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. SAE: an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience; persistent or significant disability/incapacity; congenital anomaly. MAAE: an AE leading to a non-routine/unscheduled medically-attended visit, to or from medical doctor for any reason. AESI: an event of scientific and medical interest specific to further understanding of study drug safety profile and require close monitoring and rapid communication by investigators to Sponsor.
Time Frame: During the 28-day follow-up period after vaccination (vaccines administered on Days 1 and 29 [only for primary vaccination cohort])
Population: Seronegative safety analysis set included all participants who received at least 1 dose of study treatment, were analysed according to treatment actually received, and were seronegative at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- mRNA:AZD2816
Number analyzed (Participants) | 379 | 348 | 302
Participants
  Any unsolicited TEAEs | 96 | 70 | 79
  Any TESAEs | 1 | 0 | 1
  Any MAAEs | 31 | 26 | 24
  Any AESIs | 10 | 1 | 6

3. Primary Outcome: Number of Participants With Abnormal Laboratory Parameters Reported as TEAEs in Primary Vaccination Cohort:- AZD2816 (4), Booster Cohorts:-AZD1222:AZD2816 and mRNA:AZD2816
Description: Number of participants with abnormal laboratory parameters reported as TEAEs are reported. Laboratory tests included haematology and clinical chemistry.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- mRNA:AZD2816
Number analyzed (Participants) | 379 | 348 | 302
Participants
  Anaemia | 1 | 0 | 0
  Eosinophilia | 1 | 0 | 1
  Iron deficiency anaemia | 2 | 0 | 1
  Hypercholesterolaemia | 1 | 0 | 0
  Alanine aminotransferase increased | 1 | 0 | 0
  Fibrin D dimer increased | 1 | 2 | 4
  Haematocrit decreased | 1 | 0 | 0
  Haemoglobin decreased | 2 | 0 | 0
  Transaminases increased | 1 | 0 | 0
  Lymphopenia | 0 | 1 | 0
  Normochromic normocytic anaemia | 0 | 1 | 0
  Thrombocytopenia | 0 | 1 | 0
  Hyponatraemia | 0 | 1 | 0
  Blood creatine increased | 0 | 1 | 0
  White blood cell count increased | 0 | 2 | 0
  Aspartate aminotransferase increased | 0 | 0 | 1
  Blood alkaline phosphatase increased | 0 | 0 | 1
  Blood fibrinogen increased | 0 | 0 | 2
  Vitamin D decreased | 0 | 0 | 1

4. Primary Outcome: Geometric Mean Titre (GMT) of SARS-CoV-2 Neutralizing Antibodies (nAb) Against B.1.351 Variant Elicited by Primary Vaccination Cohort:- AZD2816 (4) and the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Primary Vaccination Cohort:- AZD2816 (4) with response against B.1.351 variant is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: Seronegative immunogenicity analysis set: all participants who received at least 1 dose of study treatment, had baseline and post-dose antibody measurements, at least 1 post-dose quantifiable serum titre, and no protocol deviations judged to have potential to interfere with the antibody response, were analysed according to treatment actually received, and were seronegative at baseline. The number of participants analyzed denotes those participants who were evaluable at the specified time frame.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Groups:
- Primary Vaccination Cohort:- AZD1222 (4): Previously unvaccinated seronegative participants received IM AZD1222 5*10^10 vp on Days 1 and 29 (4-week dosing interval).
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 342 | 348
1/dilution | 790.96 [735.29 to 850.85] | 661.29 [617.16 to 708.57]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using analysis of covariance (ANCOVA); Test type: Non-Inferiority — Noninferiority was demonstrated if the lower limit of the 2-sided 95% confidence interval (CI) of the GMT ratio of the comparator group and reference group was > 0.67; GMT ratio = 1.19, 95% CI 2-sided [1.08 to 1.32]

5. Primary Outcome: GMT of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- AZD1222:AZD1222 and AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- AZD1222:AZD1222 is the comparator group and AZD1222 in Historical Control is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Groups:
- Booster Cohort:- AZD1222:AZD1222: Seronegative participants, who previously received 2 doses of AZD1222 vaccine according to the authorized dose and dosing regimen, with second dose administered at least 90 days prior to study treatment, received booster dose of IM AZD1222 5*10^10 vp on Day 1.
- Historical Control: A sub-population of participants from Study D8110C00001 (NCT04516746), who were matched with the AZD1222 cohort in this study based on age, body mass index, sex, and presence of baseline comorbidities are included and selected from those treated with 2 doses of AZD1222, gave informed consent, had no protocol deviations judged to have the potential to interfere with the generation or interpretation of an immune response, had baseline and Day 57 pseudoneutralisation data, and prior to Day 57 had no prohibited concomitant medications, Emergency Use Authorization (EUA) vaccinations, or positive polymerase chain reaction (PCR) test.
Arm/Group | Booster Cohort:- AZD1222:AZD1222 | Historical Control
Number analyzed (Participants) | 329 | 508
1/dilution | 246.45 [227.39 to 267.12] | 242.80 [224.82 to 262.23]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD1222 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — Noninferiority was demonstrated if the lower limit of the 2-sided 95% CI of the GMT ratio of the comparator group and reference group is > 0.67; GMT ratio = 1.02, 95% CI 2-sided [0.90 to 1.14]

6. Primary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against the B.1.351 Variant Elicited by Primary Vaccination Cohort:- AZD2816 (4) and the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Primary Vaccination Cohort:- AZD2816 (4) with response against B.1.351 variant is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 342 | 344
Percentage of participants | 89.47 [85.73 to 92.52] | 87.79 [83.86 to 91.06]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI rate difference in seroresponse between the comparator group and reference group was > or =-10%; Seroresponse difference = 1.68, 95% CI 2-sided [-3.11 to 6.49]

7. Primary Outcome: GMT of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- mRNA:AZD1222 and AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- mRNA:AZD1222 is the comparator group and AZD1222 in Historical Control is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Groups:
- Booster Cohort:- mRNA:AZD1222: Seronegative participants, who previously received 2 doses of approved mRNA based vaccine according to the authorized dose and dosing regimen, with second dose administered at least 90 days prior to study treatment, received booster dose of IM AZD1222 5*10^10 vp on Day 1.
- Historical Control: A sub-population of participants from Study D8110C00001 (NCT04516746), who were matched with the AZD1222 cohort in this study based on age, body mass index, sex, and presence of baseline comorbidities are included and selected from those treated with 2 doses of AZD1222, gave informed consent, had no protocol deviations judged to have the potential to interfere with the generation or interpretation of an immune response, had baseline and Day 57 pseudoneutralisation data, and prior to Day 57 had no prohibited concomitant medications, EUA vaccinations, or positive PCR test.
Arm/Group | Booster Cohort:- mRNA:AZD1222 | Historical Control
Number analyzed (Participants) | 280 | 508
1/dilution | 841.96 [790.34 to 896.96] | 242.80 [224.82 to 262.23]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD1222 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; GMT ratio = 3.47, 95% CI 2-sided [3.09 to 3.89]

8. Secondary Outcome: Number of Participants With Local and Systemic Solicited TEAEs
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. Solicited AEs are local or systemic predefined events for assessment of reactogenicity. An e-diary was used to collect information on the timing and severity of the solicited AEs. Local AEs included pain, redness/erythema, tenderness, induration/swelling at the site of the injection. Systemic AEs included fever (> 100 °F/37.8 °C), chills, muscle pains, fatigue, headache, malaise, nausea, and vomiting.
Time Frame: During the 7-day follow-up period after vaccination (vaccines administered on Days 1 and 29 or Day 85 [only for primary vaccination cohorts])
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Primary Vaccination Cohort:- AZD1222 + AZD2816 (4): Previously unvaccinated seronegative participants received IM AZD1222 5*10^10 vp on Day 1 and IM AZD2816 5*10^10 vp on Day 29 (4-week dosing interval).
- Primary Vaccination Cohort:- AZD2816 (12): Previously unvaccinated seronegative participants received IM AZD2816 5*10^10 vp on Days 1 and 85 (12-week dosing interval).
Arm/Group | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD2816 (12) | Booster Cohort:- AZD1222:AZD1222 | Booster Cohort:- mRNA:AZD1222
Number analyzed (Participants) | 373 | 188 | 340 | 299
Participants
  Any solicited AEs | 322 | 168 | 266 | 269
  Any local solicited AEs | 285 | 146 | 209 | 228
  Any systemic solicited AEs | 296 | 153 | 206 | 238

9. Secondary Outcome: Number of Participants With Unsolicited TEAEs, TESAEs, MAAEs, and AESIs
Description: as for outcome 2
Time Frame: During the 28-day follow-up period after vaccination (vaccines administered on Days 1 and 29 or Day 85 [only for primary vaccination cohorts])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD2816 (12) | Booster Cohort:- AZD1222:AZD1222 | Booster Cohort:- mRNA:AZD1222
Number analyzed (Participants) | 380 | 191 | 349 | 300
Participants
  Any unsolicited TEAEs | 93 | 67 | 81 | 73
  Any TESAEs | 2 | 0 | 0 | 0
  Any MAAEs | 37 | 25 | 34 | 16
  Any AESIs | 9 | 7 | 3 | 6

10. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Primary Vaccination Cohort:- AZD2816 (4) and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Primary Vaccination Cohort:- AZD2816 (4) is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against B.1.351 variant.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 342 | 348
1/dilution | 865.48 [837.85 to 894.02] | 269.89 [260.72 to 279.37]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — Noninferiority was demonstrated if the lower limit of the 2-sided 95% CI of the GMT ratio of the comparator group and reference group was > 0.67; GMT ratio = 3.21, 95% CI 2-sided [3.06 to 3.36]

11. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) and the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) with response against B.1.351 variant is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 334 | 348
1/dilution | 405.20 [373.64 to 439.43] | 800.92 [745.59 to 860.36]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.50, 95% CI 2-sided [0.45 to 0.56]

12. Secondary Outcome: GMT of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD2816 (4) and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Primary Vaccination Cohort:- AZD2816 (4) is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 342 | 348
1/dilution | 222.75 [201.60 to 246.12] | 719.37 [654.68 to 790.46]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.31, 95% CI 2-sided [0.27 to 0.35]

13. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- AZD1222:AZD2816 and the Original Wuhan-Hu-1 Strain Elicited by AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- AZD1222:AZD2816 with response against B.1.351 variant is the comparator group and AZD1222 in Historical Control with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- AZD1222:AZD2816 | Historical Control
Number analyzed (Participants) | 322 | 508
1/dilution | 341.96 [315.48 to 370.66] | 242.80 [224.82 to 262.23]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD2816 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 1.41, 95% CI 2-sided [1.25 to 1.58]

14. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- AZD1222:AZD2816 and Booster Cohort:- AZD1222:AZD1222
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- AZD1222:AZD2816 is the comparator group and Booster Cohort:- AZD1222:AZD1222 is the reference group, both compared for response against B.1.351 variant.
Time Frame: 28 days after booster dose (Day 29)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- AZD1222:AZD1222
Number analyzed (Participants) | 322 | 329
1/dilution | 341.96 [315.48 to 370.66] | 185.70 [169.32 to 203.66]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD2816 vs Booster Cohort:- AZD1222:AZD1222; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 1.84, 95% CI 2-sided [1.63 to 2.08]

15. Secondary Outcome: GMT of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- AZD1222:AZD2816 and AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- AZD1222:AZD2816 is the comparator group and AZD1222 in Historical Control is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- AZD1222:AZD2816 | Historical Control
Number analyzed (Participants) | 322 | 508
1/dilution | 213.26 [197.45 to 230.34] | 242.80 [224.82 to 262.23]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD2816 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.88, 95% CI 2-sided [0.78 to 0.99]

16. Secondary Outcome: GMT of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- AZD1222:AZD2816 and Booster Cohort:- AZD1222:AZD1222
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- AZD1222:AZD2816 is the comparator group and Booster Cohort:- AZD1222:AZD1222 is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: 28 days after booster dose (Day 29)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- AZD1222:AZD1222
Number analyzed (Participants) | 322 | 329
1/dilution | 213.26 [197.45 to 230.34] | 246.45 [227.39 to 267.12]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD2816 vs Booster Cohort:- AZD1222:AZD1222; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.87, 95% CI 2-sided [0.78 to 0.97]

17. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- AZD1222:AZD2816 and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- AZD1222:AZD2816 is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against B.1.351 variant.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Primary Vaccination Cohort: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Groups:
- Primary Vaccination Cohort:- AZD1222 (4): Previously unvaccinated seronegative participants received IM AZD1222 5*10^10 vp on Days 1 and 29.
Arm/Group | Booster Cohort:- AZD1222:AZD2816 | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 322 | 348
1/dilution | 341.96 [315.48 to 370.66] | 360.43 [324.90 to 399.84]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD2816 vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.95, 95% CI 2-sided [0.83 to 1.08]

18. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- mRNA:AZD2816 and the Original Wuhan-Hu-1 Strain Elicited by AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- mRNA:AZD2816 with response against B.1.351 variant is the comparator group and AZD1222 in Historical Control with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- mRNA:AZD2816 | Historical Control
Number analyzed (Participants) | 280 | 508
1/dilution | 1587.58 [1463.98 to 1721.61] | 242.80 [224.82 to 262.23]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD2816 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 6.56, 95% CI 2-sided [5.82 to 7.40]

19. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- mRNA:AZD2816 and Booster Cohort:- mRNA:AZD1222
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- mRNA:AZD2816 is the comparator group and Booster Cohort:- mRNA:AZD1222 is the reference group, both compared for response against B.1.351 variant.
Time Frame: 28 days after booster dose (Day 29)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- mRNA:AZD2816 | Booster Cohort:- mRNA:AZD1222
Number analyzed (Participants) | 280 | 280
1/dilution | 1587.58 [1463.98 to 1721.61] | 718.90 [670.46 to 770.84]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD2816 vs Booster Cohort:- mRNA:AZD1222; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 2.22, 95% CI 2-sided [1.99 to 2.47]

20. Secondary Outcome: GMT of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- mRNA:AZD2816 and AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- mRNA:AZD2816 is the comparator group and AZD1222 in Historical Control is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- mRNA:AZD2816 | Historical Control
Number analyzed (Participants) | 280 | 508
1/dilution | 1052.73 [974.55 to 1137.19] | 242.80 [224.82 to 262.23]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD2816 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; GMT ratio = 4.35, 95% CI 2-sided [3.86 to 4.90]

21. Secondary Outcome: GMT of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- mRNA:AZD2816 and Booster Cohort:- mRNA:AZD1222
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- mRNA:AZD2816 is the comparator group and Booster Cohort:- mRNA:AZD1222 is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: 28 days after booster dose (Day 29)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- mRNA:AZD2816 | Booster Cohort:- mRNA:AZD1222
Number analyzed (Participants) | 280 | 280
1/dilution | 1052.73 [974.55 to 1137.19] | 841.96 [790.34 to 896.96]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD2816 vs Booster Cohort:- mRNA:AZD1222; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 1.25, 95% CI 2-sided [1.13 to 1.39]

22. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- mRNA:AZD2816 and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- mRNA:AZD2816 is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against B.1.351 variant.
Time Frame: as for outcome 17
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- mRNA:AZD2816 | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 280 | 348
1/dilution | 1587.58 [1463.98 to 1721.61] | 360.43 [324.90 to 399.84]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD2816 vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 4.42, 95% CI 2-sided [3.85 to 5.08]

23. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- AZD1222:AZD2816 and the Original Wuhan-Hu-1 Strain Elicited by AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- AZD1222:AZD2816 with response against B.1.351 variant is the comparator group and AZD1222 in Historical Control with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- AZD1222:AZD2816 | Historical Control
Number analyzed (Participants) | 320 | 508
Percentage of participants | 82.81 [78.22 to 86.78] | 84.06 [80.58 to 87.13]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD2816 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -1.24, 95% CI 2-sided [-6.62 to 3.84]

24. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- AZD1222:AZD2816 and Booster Cohort:- AZD1222:AZD1222
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- AZD1222:AZD2816 is the comparator group and Booster Cohort:- AZD1222:AZD1222 is the reference group, both compared for response against B.1.351 variant.
Time Frame: 28 days after booster dose (Day 29)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- AZD1222:AZD1222
Number analyzed (Participants) | 320 | 329
Percentage of participants | 82.81 [78.22 to 86.78] | 65.96 [60.56 to 71.07]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD2816 vs Booster Cohort:- AZD1222:AZD1222; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 16.86, 95% CI 2-sided [10.18 to 23.32]

25. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- AZD1222:AZD2816 and AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- AZD1222:AZD2816 is the comparator group and AZD1222 in Historical Control is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- AZD1222:AZD2816 | Historical Control
Number analyzed (Participants) | 320 | 508
Percentage of participants | 65.94 [60.46 to 71.12] | 84.06 [80.58 to 87.13]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD2816 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -18.12, 95% CI 2-sided [-24.22 to -12.07]

26. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- AZD1222:AZD2816 and Booster Cohort:- AZD1222:AZD1222
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- AZD1222:AZD2816 is the comparator group and Booster Cohort:- AZD1222:AZD1222 is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: 28 days after booster dose (Day 29)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- AZD1222:AZD1222
Number analyzed (Participants) | 320 | 329
Percentage of participants | 65.94 [60.46 to 71.12] | 65.96 [60.56 to 71.07]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD2816 vs Booster Cohort:- AZD1222:AZD1222; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -0.02, 95% CI 2-sided [-7.28 to 7.23]

27. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- AZD1222:AZD2816 and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- AZD1222:AZD2816 is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against B.1.351 variant.
Time Frame: as for outcome 17
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- AZD1222:AZD2816 | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 320 | 344
Percentage of participants | 82.81 [78.22 to 86.78] | 51.45 [46.03 to 56.85]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD2816 vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 31.36, 95% CI 2-sided [24.44 to 37.82]

28. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- mRNA:AZD2816 and the Original Wuhan-Hu-1 Strain Elicited by AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- mRNA:AZD2816 with response against B.1.351 variant is the comparator group and AZD1222 in Historical Control with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- mRNA:AZD2816 | Historical Control
Number analyzed (Participants) | 277 | 508
Percentage of participants | 80.51 [75.34 to 85.00] | 84.06 [80.58 to 87.13]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD2816 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -3.55, 95% CI 2-sided [-9.40 to 1.90]

29. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- mRNA:AZD2816 and Booster Cohort:- mRNA:AZD1222
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- mRNA:AZD2816 is the comparator group and Booster Cohort:- mRNA:AZD1222 is the reference group, both compared for response against B.1.351 variant.
Time Frame: 28 days after booster dose (Day 29)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- mRNA:AZD2816 | Booster Cohort:- mRNA:AZD1222
Number analyzed (Participants) | 277 | 280
Percentage of participants | 80.51 [75.34 to 85.00] | 57.50 [51.48 to 63.36]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD2816 vs Booster Cohort:- mRNA:AZD1222; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 23.01, 95% CI 2-sided [15.41 to 30.23]

30. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- mRNA:AZD2816 and AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- mRNA:AZD2816 is the comparator group and AZD1222 in Historical Control is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- mRNA:AZD2816 | Historical Control
Number analyzed (Participants) | 277 | 508
Percentage of participants | 49.82 [43.78 to 55.86] | 84.06 [80.58 to 87.13]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD2816 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -34.24, 95% CI 2-sided [-40.77 to -27.45]

31. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- mRNA:AZD2816 and Booster Cohort:- mRNA:AZD1222
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- mRNA:AZD2816 is the comparator group and Booster Cohort:- mRNA:AZD1222 is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: 28 days after booster dose (Day 29)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- mRNA:AZD2816 | Booster Cohort:- mRNA:AZD1222
Number analyzed (Participants) | 277 | 280
Percentage of participants | 49.82 [43.78 to 55.86] | 42.86 [36.99 to 48.88]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD2816 vs Booster Cohort:- mRNA:AZD1222; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 6.96, 95% CI 2-sided [-1.31 to 15.10]

32. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- mRNA:AZD2816 and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- mRNA:AZD2816 is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against B.1.351 variant.
Time Frame: as for outcome 17
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- mRNA:AZD2816 | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 277 | 344
Percentage of participants | 80.51 [75.34 to 85.00] | 51.45 [46.03 to 56.85]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD2816 vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 29.05, 95% CI 2-sided [21.76 to 35.81]

33. Secondary Outcome: Number of Participants With TESAEs, MAAEs, and AESIs From Day 1 Through 6 Months Post Last Dose
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. The MAAEs are defined as AEs leading to medically-attended visits that were not routine visits, or an otherwise unscheduled visit to or from medical doctor for any reason. The AESIs are events of scientific and medical interest specific to the further understanding of study drug safety profile and require close monitoring and rapid communication by the investigators to the Sponsor.
Time Frame: During the 6 months follow-up period after vaccination (vaccines administered on Days 1 and 29 or Day 85 [only for primary vaccination cohorts])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD2816 (12) | Booster Cohort:- AZD1222:AZD1222 | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- mRNA:AZD1222 | Booster Cohort:- mRNA:AZD2816
Number analyzed (Participants) | 379 | 380 | 191 | 349 | 348 | 300 | 302
Participants
  Any TESAEs | 2 | 5 | 2 | 6 | 7 | 3 | 4
  Any MAAEs | 69 | 82 | 50 | 72 | 65 | 47 | 58
  Any AESIs | 48 | 51 | 32 | 41 | 42 | 31 | 33

34. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against B.1.351 variant.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 334 | 348
1/dilution | 446.63 [432.91 to 460.78] | 329.46 [319.47 to 339.76]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 1.36, 95% CI 2-sided [1.30 to 1.42]

35. Secondary Outcome: GMT of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against the Original Wuhan-Hu-1 Strain.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 334 | 348
1/dilution | 581.78 [553.12 to 611.92] | 769.03 [731.95 to 808.00]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.76, 95% CI 2-sided [0.70 to 0.81]

36. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant and the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD2816 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Primary Vaccination Cohort:- AZD2816 (4) with response against B.1.351 variant is the comparator group and Primary Vaccination Cohort:- AZD2816 (4) with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Groups:
- Primary Vaccination Cohort:- AZD2816 (4) (Comparator); Primary Vaccination Cohort:- AZD2816 (4) (Reference): Previously unvaccinated seronegative participants received IM AZD2816 5*10^10 vp on Days 1 and 29 (4-week dosing interval).
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) (Comparator) | Primary Vaccination Cohort:- AZD2816 (4) (Reference)
Number analyzed (Participants) | 342 | 342
1/dilution | 718.10 [662.58 to 778.27] | 185.70 [168.16 to 205.07]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD2816 (4) (Comparator) vs Primary Vaccination Cohort:- AZD2816 (4) (Reference); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 3.87, 95% CI 2-sided [3.40 to 4.39]

37. Secondary Outcome: GMT of SARS-CoV-2 nAb Against the B.1.351 Variant and the Original Wuhan-Hu-1 Strain by Primary Vaccination Cohort:- AZD1222 + AZD2816 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) with response against B.1.351 variant is the comparator group and Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Groups:
- Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (Comparator); Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (Reference): Previously unvaccinated seronegative participants received IM AZD1222 5*10^10 vp on Day 1 and IM AZD2816 5*10^10 vp on Day 29 (4-week dosing interval).
Arm/Group | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (Comparator) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (Reference)
Number analyzed (Participants) | 334 | 334
1/dilution | 392.13 [380.34 to 404.28] | 586.00 [566.15 to 606.54]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (Comparator) vs Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (Reference); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.67, 95% CI 2-sided [0.64 to 0.70]

38. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Primary Vaccination Cohort:- AZD2816 (4) and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Primary Vaccination Cohort:- AZD2816 (4) is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against B.1.351 variant.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 342 | 344
Percentage of participants | 100 [98.73 to NA] — Upper limit of 95% confidence interval was not evaluable as all participants had seroresponse. | 99.42 [97.92 to 99.93]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 0.58, 95% CI 2-sided [-0.61 to 2.09]

39. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD2816 (4) and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Primary Vaccination Cohort:- AZD2816 (4) is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 342 | 344
Percentage of participants | 49.42 [44.00 to 54.85] | 84.59 [80.34 to 88.24]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -35.18, 95% CI 2-sided [-41.46 to -28.44]

40. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) and the Original Wuhan Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) with response against B.1.351 variant is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 334 | 344
Percentage of participants | 62.57 [57.14 to 67.78] | 87.50 [83.53 to 90.80]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -24.93, 95% CI 2-sided [-31.06 to -18.56]

41. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against B.1.351 variant.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 334 | 344
Percentage of participants | 99.40 [97.85 to 99.93] | 99.42 [97.92 to 99.93]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -0.02, 95% CI 2-sided [-1.63 to 1.56]

42. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 334 | 344
Percentage of participants | 80.24 [75.56 to 84.38] | 99.42 [97.92 to 99.93]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -19.18, 95% CI 2-sided [-23.80 to -14.98]

43. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant and the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD2816 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Primary Vaccination Cohort:- AZD2816 (4) with response against B.1.351 variant is the comparator group and Primary Vaccination Cohort:- AZD2816 (4) with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) (Comparator) | Primary Vaccination Cohort:- AZD2816 (4) (Reference)
Number analyzed (Participants) | 342 | 342
Percentage of participants | 88.60 [84.74 to 91.76] | 49.42 [44.00 to 54.85]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD2816 (4) (Comparator) vs Primary Vaccination Cohort:- AZD2816 (4) (Reference); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 39.18, 95% CI 2-sided [32.68 to 45.21]

44. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant and the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD1222 + AZD2816 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) with response against B.1.351 variant is the comparator group and Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (Comparator) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (Reference)
Number analyzed (Participants) | 334 | 334
Percentage of participants | 99.40 [97.85 to 99.93] | 99.40 [97.85 to 99.93]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (Comparator) vs Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (Reference); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 0.00, 95% CI 2-sided [-1.62 to 1.62]

45. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- AZD1222:AZD1222 and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- AZD1222:AZD1222 is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against B.1.351 variant.
Time Frame: as for outcome 17
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- AZD1222:AZD1222 | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 329 | 348
1/dilution | 185.70 [169.32 to 203.66] | 360.43 [324.90 to 399.84]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD1222 vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.52, 95% CI 2-sided [0.45 to 0.59]

46. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- AZD1222:AZD1222 and the Original Wuhan-Hu-1 Strain Elicited by AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- AZD1222:AZD1222 with response against B.1.351 variant is the comparator group and AZD1222 in Historical Control with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- AZD1222:AZD1222 | Historical Control
Number analyzed (Participants) | 329 | 508
1/dilution | 185.70 [169.32 to 203.66] | 242.80 [224.82 to 262.23]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD1222 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.76, 95% CI 2-sided [0.68 to 0.86]

47. Secondary Outcome: GMT of SARS-CoV-2 nAb Against the B.1.351 Variant and the Original Wuhan-Hu-1 Strain by Booster Cohort:- AZD1222:AZD2816
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- AZD1222:AZD2816 with response against B.1.351 variant is the comparator group and Booster Cohort:- AZD1222:AZD2816 with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Groups:
- Booster Cohort:- AZD1222:AZD2816 (Comparator); Booster Cohort:- AZD1222:AZD2816 (Reference): Seronegative participants, who previously received 2 doses of AZD1222 vaccine according to the authorized dose and dosing regimen, with second dose administered at least 90 days prior to study treatment, received booster dose of IM AZD2816 5*10^10 vp on Day 1.
Arm/Group | Booster Cohort:- AZD1222:AZD2816 (Comparator) | Booster Cohort:- AZD1222:AZD2816 (Reference)
Number analyzed (Participants) | 322 | 322
1/dilution | 341.96 [315.48 to 370.66] | 213.26 [197.45 to 230.34]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD2816 (Comparator) vs Booster Cohort:- AZD1222:AZD2816 (Reference); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 1.60, 95% CI 2-sided [1.43 to 1.79]

48. Secondary Outcome: GMT of SARS-CoV-2 nAb Against the B.1.351 Variant and the Original Wuhan-Hu-1 Strain by Booster Cohort:- AZD1222:AZD1222
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information.Booster Cohort:- AZD1222:AZD1222 with response against B.1.351 variant is the comparator group and Booster Cohort:- AZD1222:AZD1222 with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Groups:
- Booster Cohort:- AZD1222:AZD1222 (Comparator); Booster Cohort:- AZD1222:AZD1222 (Reference): Seronegative participants, who previously received 2 doses of AZD1222 vaccine according to the authorized dose and dosing regimen, with second dose administered at least 90 days prior to study treatment, received booster dose of IM AZD1222 5*10^10 vp on Day 1.
Arm/Group | Booster Cohort:- AZD1222:AZD1222 (Comparator) | Booster Cohort:- AZD1222:AZD1222 (Reference)
Number analyzed (Participants) | 329 | 329
1/dilution | 185.70 [169.32 to 203.66] | 246.45 [227.39 to 267.12]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD1222 (Comparator) vs Booster Cohort:- AZD1222:AZD1222 (Reference); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.75, 95% CI 2-sided [0.67 to 0.85]

49. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- AZD1222:AZD1222 and AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- AZD1222:AZD1222 is the comparator group and AZD1222 in Historical Control is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- AZD1222:AZD1222 | Historical Control
Number analyzed (Participants) | 329 | 508
Percentage of participants | 65.96 [60.56 to 71.07] | 84.06 [80.58 to 87.13]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD1222 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -18.10, 95% CI 2-sided [-24.13 to -12.10]

50. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- AZD1222:AZD1222 and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- AZD1222:AZD1222 is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against B.1.351 Variant.
Time Frame: as for outcome 17
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- AZD1222:AZD1222 | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 329 | 344
Percentage of participants | 65.96 [60.56 to 71.07] | 51.45 [46.03 to 56.85]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD1222 vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 14.50, 95% CI 2-sided [7.07 to 21.71]

51. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- AZD1222:AZD1222 and the Original Wuhan-Hu-1 Strain Elicited by AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- AZD1222:AZD1222 with response against B.1.351 variant is the comparator group and AZD1222 in Historical Control with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- AZD1222:AZD1222 | Historical Control
Number analyzed (Participants) | 329 | 508
Percentage of participants | 65.96 [60.56 to 71.07] | 84.06 [80.58 to 87.13]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD1222 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -18.10, 95% CI 2-sided [-24.13 to -12.10]

52. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant and the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- AZD1222:AZD2816
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- AZD1222:AZD2816 with response against B.1.351 variant is the comparator group and Booster Cohort:- AZD1222:AZD2816 with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- AZD1222:AZD2816 (Comparator) | Booster Cohort:- AZD1222:AZD2816 (Reference)
Number analyzed (Participants) | 320 | 320
Percentage of participants | 82.81 [78.22 to 86.78] | 65.94 [60.46 to 71.12]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD2816 (Comparator) vs Booster Cohort:- AZD1222:AZD2816 (Reference); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 16.87, 95% CI 2-sided [10.15 to 23.40]

53. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant and the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- AZD1222:AZD1222
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- AZD1222:AZD1222 with response against B.1.351 variant is the comparator group and Booster Cohort:- AZD1222:AZD1222 with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- AZD1222:AZD1222 (Comparator) | Booster Cohort:- AZD1222:AZD1222 (Reference)
Number analyzed (Participants) | 329 | 329
Percentage of participants | 65.96 [60.56 to 71.07] | 65.96 [60.56 to 71.07]
Statistical Analysis 1: Comparison: Booster Cohort:- AZD1222:AZD1222 (Comparator) vs Booster Cohort:- AZD1222:AZD1222 (Reference); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 0.00, 95% CI 2-sided [-7.21 to 7.21]

54. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- mRNA:AZD1222 and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- mRNA:AZD1222 is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against B.1.351 variant.
Time Frame: as for outcome 17
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- mRNA:AZD1222 | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 280 | 348
1/dilution | 718.90 [670.46 to 770.84] | 360.43 [324.90 to 399.84]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD1222 vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 2.00, 95% CI 2-sided [1.75 to 2.28]

55. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- mRNA:AZD1222 and the Original Wuhan-Hu-1 Strain Elicited by AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- mRNA:AZD1222 with response against B.1.351 variant is the comparator group and AZD1222 in Historical Control with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Booster Cohort:- mRNA:AZD1222 | Historical Control
Number analyzed (Participants) | 280 | 508
1/dilution | 718.90 [670.46 to 770.84] | 242.80 [224.82 to 262.23]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD1222 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 2.96, 95% CI 2-sided [2.64 to 3.32]

56. Secondary Outcome: GMT of SARS-CoV-2 nAb Against the B.1.351 Variant and the Original Wuhan-Hu-1 Strain by Booster Cohort:- mRNA:AZD2816
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- mRNA:AZD2816 with response against B.1.351 variant is the comparator group and Booster Cohort:- mRNA:AZD2816 with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Groups:
- Booster Cohort:- mRNA:AZD2816 (Comparator); Booster Cohort:- mRNA:AZD2816 (Reference): Seronegative participants, who previously received 2 doses of approved mRNA based vaccine according to the authorized dose and dosing regimen, with second dose administered at least 90 days prior to study treatment, received booster dose of IM AZD2816 5*10^10 vp on Day 1.
Arm/Group | Booster Cohort:- mRNA:AZD2816 (Comparator) | Booster Cohort:- mRNA:AZD2816 (Reference)
Number analyzed (Participants) | 280 | 280
1/dilution | 1587.58 [1463.98 to 1721.61] | 1052.73 [974.55 to 1137.19]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD2816 (Comparator) vs Booster Cohort:- mRNA:AZD2816 (Reference); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 1.51, 95% CI 2-sided [1.35 to 1.69]

57. Secondary Outcome: GMT of SARS-CoV-2 nAb Against the B.1.351 Variant and the Original Wuhan-Hu-1 Strain by Booster Cohort:- mRNA:AZD1222
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Booster Cohort:- mRNA:AZD1222 with response against B.1.351 variant is the comparator group and Booster Cohort:- mRNA:AZD1222 with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Groups:
- Booster Cohort:- mRNA:AZD1222 (Comparator); Booster Cohort:- mRNA:AZD1222 (Reference): Seronegative participants, who previously received 2 doses of approved mRNA based vaccine according to the authorized dose and dosing regimen, with second dose administered at least 90 days prior to study treatment, received booster dose of IM AZD1222 5*10^10 vp on Day 1.
Arm/Group | Booster Cohort:- mRNA:AZD1222 (Comparator) | Booster Cohort:- mRNA:AZD1222 (Reference)
Number analyzed (Participants) | 280 | 280
1/dilution | 718.90 [670.46 to 770.84] | 841.96 [790.34 to 896.96]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD1222 (Comparator) vs Booster Cohort:- mRNA:AZD1222 (Reference); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.85, 95% CI 2-sided [0.78 to 0.94]

58. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- mRNA:AZD1222 and AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- mRNA:AZD1222 is the comparator group and AZD1222 in Historical Control is the reference group, both compared for response against the original Wuhan-Hu-1 strain.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- mRNA:AZD1222 | Historical Control
Number analyzed (Participants) | 280 | 508
Percentage of participants | 42.86 [36.99 to 48.88] | 84.06 [80.58 to 87.13]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD1222 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -41.20, 95% CI 2-sided [-47.57 to -34.41]

59. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- mRNA:AZD1222 and Primary Vaccination Cohort:- AZD1222 (4)
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- mRNA:AZD1222 is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) is the reference group, both compared for response against B.1.351 Variant.
Time Frame: as for outcome 17
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- mRNA:AZD1222 | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 280 | 344
Percentage of participants | 57.50 [51.48 to 63.36] | 51.45 [46.03 to 56.85]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD1222 vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 6.05, 95% CI 2-sided [-1.81 to 13.77]

60. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Booster Cohort:- mRNA:AZD1222 and the Original Wuhan-Hu-1 Strain Elicited by AZD1222 in Historical Control
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- mRNA:AZD1222 with response against B.1.351 variant is the comparator group and AZD1222 in Historical Control with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: Booster Cohort: 28 days after booster dose (Day 29) and Historical Control: 28 days after the second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- mRNA:AZD1222 | Historical Control
Number analyzed (Participants) | 280 | 508
Percentage of participants | 57.50 [51.48 to 63.36] | 84.06 [80.58 to 87.13]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD1222 vs Historical Control; The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = -26.56, 95% CI 2-sided [-33.10 to -19.94]

61. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant and the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- mRNA:AZD2816
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- mRNA:AZD2816 with response against B.1.351 variant is the comparator group and Booster Cohort:- mRNA:AZD2816 with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- mRNA:AZD2816 (Comparator) | Booster Cohort:- mRNA:AZD2816 (Reference)
Number analyzed (Participants) | 277 | 277
Percentage of participants | 80.51 [75.34 to 85.00] | 49.82 [43.78 to 55.86]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD2816 (Comparator) vs Booster Cohort:- mRNA:AZD2816 (Reference); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 30.69, 95% CI 2-sided [22.94 to 37.90]

62. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 nAb Against B.1.351 Variant and the Original Wuhan-Hu-1 Strain Elicited by Booster Cohort:- mRNA:AZD1222
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline. Booster Cohort:- mRNA:AZD1222 with response against B.1.351 variant is the comparator group and Booster Cohort:- mRNA:AZD1222 with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after second dose (Day 57)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Booster Cohort:- mRNA:AZD1222 (Comparator) | Booster Cohort:- mRNA:AZD1222 (Reference)
Number analyzed (Participants) | 280 | 280
Percentage of participants | 57.50 [51.48 to 63.36] | 42.86 [36.99 to 48.88]
Statistical Analysis 1: Comparison: Booster Cohort:- mRNA:AZD1222 (Comparator) vs Booster Cohort:- mRNA:AZD1222 (Reference); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; Seroresponse difference = 14.64, 95% CI 2-sided [6.36 to 22.64]

63. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Primary Vaccination Cohort:- AZD2816 (4) and the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD1222 (4) on Day 29
Description: Severe acute respiratory syndrome-coronavirus-2 nAb were measured by pseudoneutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information. Primary Vaccination Cohort:- AZD2816 (4) with response against B.1.351 variant is the comparator group and Primary Vaccination Cohort:- AZD1222 (4) with response against the original Wuhan-Hu-1 strain is the reference group.
Time Frame: 28 days after first dose (Day 29)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 357 | 361
1/dilution | 364.20 [330.75 to 401.04] | 433.42 [398.43 to 471.48]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using analysis of covariance (ANCOVA); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; GMT ratio = 0.84, 95% CI 2-sided [0.74 to 0.96]

64. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Primary Vaccination Cohort:- AZD2816 (4) and Primary Vaccination Cohort:- AZD1222 (4) on Day 29
Description: as for outcome 10
Time Frame: 28 days after first dose (Day 29)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 357 | 361
1/dilution | 398.60 [381.99 to 415.95] | 233.65 [226.02 to 241.54]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 1.71, 95% CI 2-sided [1.62 to 1.80]

65. Secondary Outcome: GMT of SARS-CoV-2 nAb Against B.1.351 Variant Elicited by Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) and the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD1222 (4) on Day 29
Description: as for outcome 11
Time Frame: 28 days after first dose (Day 29)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 357 | 361
1/dilution | 261.55 [240.05 to 284.97] | 525.20 [481.75 to 572.58]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.50, 95% CI 2-sided [0.44 to 0.56]

66. Secondary Outcome: GMT of SARS-CoV-2 nAb Against the Original Wuhan-Hu-1 Strain Elicited by Primary Vaccination Cohort:- AZD2816 (4) and Primary Vaccination Cohort:- AZD1222 (4) on Day 29
Description: as for outcome 12
Time Frame: 28 days after first dose (Day 29)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 (4)
Number analyzed (Participants) | 357 | 361
1/dilution | 177.02 [160.25 to 195.53] | 471.69 [420.91 to 528.59]
Statistical Analysis 1: Comparison: Primary Vaccination Cohort:- AZD2816 (4) vs Primary Vaccination Cohort:- AZD1222 (4); The analyses were derived using ANCOVA; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMT ratio = 0.38, 95% CI 2-sided [0.32 to 0.44]

67. Secondary Outcome: GMT of ChAdOx1 nAb in Primary Vaccination Cohorts and Following a Booster Dose of AZD2816
Description: Chimpanzee adenovirus Ox1 (ChAdOx1) vector nAb were measured by neutralisation assay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information.
Time Frame: Booster Cohorts: 28 days after booster dose (Day 29) and Primary Vaccination Cohorts: 28 days after the second dose (Day 57 for 4-week dosing interval cohorts and Day 113 for 12-week dosing interval cohort)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Primary Vaccination Cohort:- AZD1222 (4) | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD2816 (12) | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- mRNA:AZD2816
Number analyzed (Participants) | 232 | 225 | 217 | 7 | 320 | 277
1/dilution | 2369.38 [2165.69 to 2592.23] | 1640.99 [1510.43 to 1782.83] | 1656.53 [1529.80 to 1793.75] | 2082.82 [787.88 to 5506.10] | 3830.85 [3574.28 to 4105.83] | 811.44 [721.11 to 913.08]

68. Secondary Outcome: Percentage of Participants With Seroresponse of ChAdOx1 nAb in Primary Vaccination Cohorts and Following a Booster Dose of AZD2816
Description: Chimpanzee adenovirus Ox1 vector nAb were measured by neutralisation assay. Seroresponse was defined as >= 4-fold increase in the GMT of nAb from baseline.
Time Frame: as for outcome 67
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Primary Vaccination Cohort:- AZD1222 (4) | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD2816 (12) | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- mRNA:AZD2816
Number analyzed (Participants) | 227 | 224 | 209 | 7 | 319 | 275
Percentage of participants | 89.43 [84.68 to 93.11] | 93.30 [89.20 to 96.20] | 91.39 [86.73 to 94.82] | 85.71 [42.13 to 99.64] | 62.07 [56.50 to 67.42] | 87.64 [83.15 to 91.28]

69. Secondary Outcome: GMT of SARS-CoV-2 Spike Protein Binding Antibodies in Primary Vaccination Cohorts and Booster Cohorts
Description: Severe acute respiratory syndrome-coronavirus-2 spike protein binding antibodies were measured by multiplexed immunoassay. The GMT was calculated as the antilogarithm of Σ(log base 2 transformed titre/n), i.e. as the anti-logarithm transformation of the mean of the log-transformed titre, where 'n' was the number of participants with titre information.
Time Frame: as for outcome 67
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | Primary Vaccination Cohort:- AZD1222 (4) | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD2816 (12) | Booster Cohort:- AZD1222:AZD1222 | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- mRNA:AZD1222 | Booster Cohort:- mRNA:AZD2816
Number analyzed (Participants) | 347 | 341 | 333 | 157 | 329 | 320 | 279 | 279
1/dilution
  B.1.351 | 28618.30 [25758.25 to 31795.92] | 29325.20 [26677.38 to 32235.81] | 23119.62 [20524.01 to 26043.50] | 43047.62 [37018.88 to 50058.17] | 14382.37 [13365.31 to 15476.82] | 16561.93 [15630.53 to 17548.83] | 45587.11 [42653.03 to 48723.02] | 65705.69 [62446.19 to 69135.33]
  Wuhan-Hu-1 | 59332.38 [53222.73 to 66143.39] | 21570.78 [19701.94 to 23616.89] | 38145.52 [33713.61 to 43160.03] | 25672.89 [21953.82 to 30021.99] | 34214.45 [31691.34 to 36938.43] | 29254.7 [27650.20 to 30952.30] | 106061.18 [98649.55 to 114029.66] | 113358.29 [107769.93 to 119236.43]

70. Secondary Outcome: Percentage of Participants With Seroresponse of SARS-CoV-2 Spike Protein Binding Antibodies in Primary Vaccination Cohorts and Booster Cohorts
Description: Severe acute respiratory syndrome-coronavirus-2 spike protein binding antibodies were measured by multiplexed immunoassay. Seroresponse was defined as >= 4-fold increase in the GMT of spike protein binding antibodies from baseline.
Time Frame: as for outcome 67
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Primary Vaccination Cohort:- AZD1222 (4) | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD2816 (12) | Booster Cohort:- AZD1222:AZD1222 | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- mRNA:AZD1222 | Booster Cohort:- mRNA:AZD2816
Number analyzed (Participants) | 345 | 341 | 333 | 156 | 329 | 320 | 279 | 278
Percentage of participants
  B.1.351 | 97.10 [94.73 to 98.60] | 97.36 [95.05 to 98.79] | 93.99 [90.88 to 96.29] | 98.08 [94.48 to 99.60] | 70.82 [65.58 to 75.68] | 75.94 [70.87 to 80.52] | 30.47 [25.12 to 36.23] | 51.08 [45.04 to 57.10]
  Wuhan-Hu-1 | 97.68 [95.48 to 98.99] | 95.01 [92.14 to 97.07] | 94.29 [91.23 to 96.53] | 96.15 [91.82 to 98.58] | 67.78 [62.44 to 72.80] | 64.69 [59.18 to 69.92] | 36.56 [30.90 to 42.51] | 41.01 [35.17 to 47.04]

71. Secondary Outcome: Correlation Between ChAdOx1 nAb and SARS-CoV-2 nAb Titres
Description: Severe acute respiratory syndrome-coronavirus-2 nAb and ChAdOx1 vector nAb were measured by pseudoneutralisation assay. Correlations were based on log2 titre values and assessed by using Spearman rank correlation for all cohorts except Primary Vaccination Cohort:- AZD2816 (12) for which Pearson correlation was used. The correlation coefficient is reported in values from +1 to -1 (+1= perfect association, 0 = no association, and -1= perfect negative association). The closer the correlation coefficient is to zero, weaker the association.
Time Frame: as for outcome 67
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | Primary Vaccination Cohort:- AZD1222 (4) | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD2816 (12) | Booster Cohort:- AZD1222:AZD1222 | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- mRNA:AZD1222 | Booster Cohort:- mRNA:AZD2816
Number analyzed (Participants) | 232 | 225 | 217 | 7 | 327 | 320 | 275 | 277
Correlation coefficient
  B.1.351 | -0.1656 [-0.29 to -0.04] | -0.0536 [-0.18 to 0.08] | -0.0783 [-0.21 to 0.06] | 0.0253 [-0.74 to 0.76] | 0.2061 [0.10 to 0.31] | 0.2297 [0.12 to 33] | 0.0225 [-0.10 to 0.14] | -0.0591 [-0.18 to 0.06]
  Wuhan-Hu-1 | -0.1263 [-0.25 to 0.00] | 0.0006 [-0.13 to 0.13] | -0.0162 [-0.15 to 0.12] | -0.1460 [-0.81 to 0.69] | 0.1288 [0.02 to 0.23] | 0.1583 [0.05 to 0.26] | 0.0005 [-0.12 to 0.12] | -0.0534 [-0.17 to 0.06]

ADVERSE EVENTS:
Time Frame: During the 6 months follow-up period after vaccination (vaccines administered on Days 1 and 29 or Day 85 [only for primary vaccination cohorts])
Description: Safety analysis set included all participants who received at least 1 dose of study treatment and were analyzed according to the treatment actually received.
Arm/Group | Primary Vaccination Cohort:- AZD1222 (4) | Primary Vaccination Cohort:- AZD2816 (4) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) | Primary Vaccination Cohort:- AZD2816 (12) | Booster Cohort:- AZD1222:AZD1222 | Booster Cohort:- AZD1222:AZD2816 | Booster Cohort:- mRNA:AZD1222 | Booster Cohort:- mRNA:AZD2816
All-Cause Mortality (participants affected / at risk) | 1/409 | 0/413 | 0/411 | 0/208 | 0/373 | 1/375 | 0/322 | 0/323
Serious Adverse Events (participants affected / at risk) | 3/409 | 3/413 | 5/411 | 2/208 | 6/373 | 8/375 | 3/322 | 5/323
Other Adverse Events (participants affected / at risk) | 32/409 | 42/413 | 42/411 | 30/208 | 39/373 | 37/375 | 25/322 | 27/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Vaccination Cohort:- AZD1222 (4) (N=409) | Primary Vaccination Cohort:- AZD2816 (4) (N=413) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (N=411) | Primary Vaccination Cohort:- AZD2816 (12) (N=208) | Booster Cohort:- AZD1222:AZD1222 (N=373) | Booster Cohort:- AZD1222:AZD2816 (N=375) | Booster Cohort:- mRNA:AZD1222 (N=322) | Booster Cohort:- mRNA:AZD2816 (N=323)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymph node tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglossal nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Vaccination Cohort:- AZD1222 (4) (N=409) | Primary Vaccination Cohort:- AZD2816 (4) (N=413) | Primary Vaccination Cohort:- AZD1222 + AZD2816 (4) (N=411) | Primary Vaccination Cohort:- AZD2816 (12) (N=208) | Booster Cohort:- AZD1222:AZD1222 (N=373) | Booster Cohort:- AZD1222:AZD2816 (N=375) | Booster Cohort:- mRNA:AZD1222 (N=322) | Booster Cohort:- mRNA:AZD2816 (N=323)
COVID-19 (Infections and infestations) | 32 (32) | 42 (42) | 42 (42) | 30 (30) | 39 (39) | 37 (37) | 25 (26) | 27 (27)

LIMITATIONS AND CAVEATS:
Since different assays were used between strains and also within the same strains between this study and historical control study D8110C00001 (NCT04516746), spike protein binding antibody results were summarised descriptively; no comparative analyses were conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2021-10-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT04973449/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT04973449/SAP_001.pdf